CLINICAL TRIAL: NCT07187947
Title: Cardiovascular Health of Transgender Individuals During the Clinical Gender-affirming Pathway
Brief Title: Cardiovascular Health of Transgender Individuals During the Gender-affirming Pathway
Acronym: CV-TGD
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Maria Cristina Meriggiola, MD, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: CV-TGD
Record Dates: First submitted 2025-08-29; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-07

CONDITIONS: Gender Incongruence; Cardiovascular (CV) Risk; Cardiovascular Disease Risk Factor; Cardiovascular Disease Acute; Cardiovascular Health Status; Cardiovascular Disease (CVD); Cardiovascular Disease Prevention
Keywords: cardiovascular risk; transgender; GAHT; GAS; hormones
MeSH Terms: conditions — Gender Dysphoria; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- AMAB: Individuals assigned male at birth, who will take on feminising gender-affirming care (i.e. cyproterone acetate/leuprorelin/triptorelin + estradiol/estradiol valerate, or estradiol/estradiol valerate alone after undergoing orchiectomy).
  Interventions: Drug: Feminizing GAHT
- AFAB: Individuals assigned male at birth, who will take on masculinizing gender-affirming care (i.e. testosterone, either before and after the hysterectomy with our without oophorectomy, if desired).
  Interventions: Drug: Masculinizing GAHT

INTERVENTIONS:
Drug: Feminizing GAHT — Before gender-affirming surgery, the regimen consists of an antiandrogen (cyproterone acetate or leuprorelin or triptorelin) plus estradiol (estradiol or estradiol valerate), whereas after an oophorectomy, estradiol/estradiol valerate can be administered alone.
  Groups: AMAB
Drug: Masculinizing GAHT — Before and after gender-affirming surgery, the regimen consists of the administration of testosterone or its esters (testosterone undecanoate, testosterone enanthate)
  Groups: AFAB

SUMMARY:
Gender incongruence, now classified in ICD-11 as a "marked and persistent incongruence between an individual's experienced gender and the gender assigned at birth," is managed in dedicated, multidisciplinary centres that coordinate psychological support with medical-surgical care.

Gender-affirming hormone therapy (GAHT) is central to this care pathway. In particular, masculinising GAHT for people assigned female at birth (AFAB) relies mainly on testosterone, and feminising or demasculinising GAHT for people assigned male at birth (AMAB) combines oestradiol with androgen-lowering agents such as cyproterone acetate or GnRH analogues (triptorelin, leuprorelin). In addition, Gender-affirming surgery (GAS) offers further individualised options: "Top" procedures- chest masculinisation for AFAB or breast augmentation for AMAB, and "Bottom" procedures** such as hysterectomy with or without oophorectomy, phalloplasty or metoidioplasty for AFAB; orchiectomy or vaginoplasty for AMAB. Other ancillary interventions include facial feminisation or voice surgery.

GAHT aims to suppress endogenous sex-hormone levels and secondary sex characteristics while inducing those consistent with the affirmed gender. Despite its widespread use, cardiovascular (CV) safety data are scant and largely observational. Sex-steroid receptors are ubiquitous in the vasculature and contribute to the sex-dimorphic patterns of CV risk seen in cisgender populations; GAHT is therefore biologically plausible as a modifier of CV outcomes in transgender people, yet robust evidence remains limited.

Current literature suggests that AFAB individuals on testosterone exhibit an up to 2.66-fold higher composite CV risk than cisgender AFAB comparators. The most consistent changes are higher blood pressure and lower HDL cholesterol; clinically significant polycythaemia is uncommon and treatable. Instead, AMAB individuals on feminising therapy do not show a clearly increased overall CV risk compared with cisgender AMAB peers, though data are inconsistent. An observational study reported that within four months of GAHT initiation, systolic blood pressure rose by 2.6 mmHg in trans men and fell by 4 mmHg in trans women, with no diastolic change in either group.

The current evidence base is weakened by small cohorts, inadequate control groups, and reliance on surrogate biochemical markers rather than hard clinical endpoints. Many studies also overlook GAHT exposure altogether, hampering meaningful interpretation. Moreover, social determinants-mental-health burden, substance use, and healthcare inequities-compound CV risk but are seldom accounted for.

Key unanswered questions include the long-term CV effects of GAHT, age-specific interactions with blood pressure and lipids, optimal therapeutic targets, and underlying mechanisms. Addressing these gaps demands rigorously designed, large-scale, prospective studies that actively involve transgender participants.

In summary, while GAHT is indispensable for gender affirmation, its cardiovascular implications-especially for AFAB individuals-warrant caution and systematic monitoring. Future evidence should inform tailored protocols that balance gender-affirming benefits against potential CV risks and integrate biomedical parameters with the broader social context impacting transgender health.

DETAILED DESCRIPTION:
Gender incongruence, described in the eleventh revision of the International Classification of Diseases (ICD-11) as "a marked and persistent incongruence between an individual's experienced gender and the gender assigned at birth" , is usually managed in specialised, multidisciplinary centres where psychologists, endocrinologists, gynaecologists, urologists and other professionals guide each person through the process of gender affirmation. Central to this pathway is gender-affirming hormone therapy (GAHT). In individuals assigned female at birth (AFAB) who seek masculinisation, treatment relies primarily on testosterone, whereas in those assigned male at birth (AMAB) who desire feminisation or demasculinisation, androgen-lowering agents such as cyproterone acetate or gonadotropin-releasing-hormone analogues (triptorelin or leuprorelin acetate) are combined with oestradiol; when complete feminisation is requested, suppression of endogenous testosterone and administration of oestradiol proceed in tandem. Gender-affirming surgery (GAS) offers further individualised possibilities: chest masculinisation in AFAB people and breast augmentation in AMAB people, orchiectomy or vaginoplasty for AMAB individuals, and hysterectomy with or without salpingo-oophorectomy followed by phalloplasty or metoidioplasty for AFAB individuals. Ancillary procedures, including facial feminisation and thyroplasty, may refine the outcome for AMAB clients.

The physiological goal of GAHT is to suppress endogenous sex-hormone levels and associated secondary sexual characteristics of the birth sex while inducing and maintaining hormone levels, and thus features, congruent with the individual's affirmed gender. Although GAHT is widely used, robust data on its cardiovascular safety remain scarce. Sex-steroid receptors are ubiquitous in vascular tissues and help explain the sex-specific patterns of cardiovascular (CV) risk seen in cisgender populations; accordingly, GAHT is biologically plausible as a modulator of CV outcomes in transgender people, yet the evidence base is still limited. Current literature points to an increased composite CV risk-up to 2.66-fold-among AFAB individuals receiving testosterone compared with cisgender AFAB controls. The most frequently reported risk-factor shifts in this group include higher blood pressure and lower high-density lipoprotein cholesterol, whereas clinically significant polycythaemia remains uncommon and treatable. By contrast, studies have not shown a statistically significant overall CV risk elevation in AMAB individuals treated with feminising regimens when compared with cisgender AMAB peers, though findings are inconsistent. One observational investigation documented that within four months of starting GAHT systolic blood pressure rose by 2.6 mmHg in trans men but fell by 4 mmHg in trans women, with diastolic values remaining unchanged in both cohorts.

Interpretation of these data is hindered by small sample sizes, the paucity of large prospective cohorts, inadequate control populations and the predominance of surrogate biochemical markers in place of clinical CV end-points. Moreover, several published studies neglect to register GAHT exposure, despite its fundamental role in transgender health management, underscoring the need for further research into the therapy's effects and risks. Social determinants of health compound the picture: higher prevalences of mental-health disorders, substance misuse and structural healthcare inequities are increasingly recognised in transgender communities and likely contribute to the observed CV risk burden.

Many critical questions therefore remain unanswered. The long-term impact of GAHT on cardiovascular morbidity and mortality is unknown, as is the extent to which a person's age modifies GAHT-related shifts in blood pressure, lipid profile or other risk parameters. Clinicians lack evidence-based targets for blood pressure or surrogate CV markers in trans men and trans women, and the biological mechanisms that underlie GAHT-related alterations in CV risk factors are not fully understood. Addressing these uncertainties will demand rigorously designed, large-scale prospective studies, conducted with active involvement of transgender participants, that integrate biomedical outcomes with the broader social realities shaping transgender health.

In summary, although GAHT is indispensable for many individuals seeking gender affirmation, its cardiovascular implications-particularly the elevated risk signalled in AFAB people receiving testosterone-warrant cautious, evidence-based monitoring. Future work should clarify long-term outcomes, refine management protocols and ensure that clinical guidelines reflect both the physiological effects of hormone therapy and the social determinants that influence cardiovascular health in transgender populations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of gender incongruence
* Age 18 years or older at the start of therapy
* Undergoing gender-affirming (replacement or suppressive) hormone therapy with testosterone or with estradiol plus anti-androgens for at least 12 months
* Provision of informed consent for study participation and for the processing of personal and sensitive data

Exclusion Criteria:

* Any hormone therapy received before recruitment
* History of cardiovascular events prior to the initiation of hormone therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Transgender AFAB and AMAB individuals diagnosed with gender incongruence who received medical therapy between January 2000 and December 2027 at the Gynecology and Reproductive Physiology Unit of the IRCCS AOU Bologna, Sant'Orsola University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Modification of vital signs | From baseline through study completion, estimated to be in 2035.
  Describe, in AFAB and AMAB transgender individuals who have been receiving gender-affirming hormone therapy (GAHT) for at least one year, changes in the following indicators of cardiovascular health: systolic BP (mmHg), diastolic BP (mmHg), mean arterial pressure (mmHg), heart rate (bpm).
Modifications in anthropometric parameters | From baseline through study completion, estimated to be in 2035.
  Describe, in AFAB and AMAB transgender individuals who have been receiving gender-affirming hormone therapy (GAHT) for at least one year, changes in the following indicators of cardiovascular health: waist (cm), hip (cm) circumference.
Modifications in blood tests | From baseline through study completion, estimated to be in 2035.
  Describe, in AFAB and AMAB transgender individuals who have been receiving gender-affirming hormone therapy (GAHT) for at least one year, changes in the following indicators of cardiovascular health:hemoglobin (g/dL), hematocrit (%), fibrinogen (mg/dL), PT (INR), aPTT (ratio), fasting glucose (mg/dL), insulin (µIU/mL), AST/ALT (U/L), total/LDL/HDL cholesterol (mg/dL), triglycerides (mg/dL), sodium/potassium (mmol/L), uric acid (mg/dL), creatinine (mg/dL), FSH/LH (IU/L), estradiol (pg/mL), testosterone (ng/dL), progesterone (ng/mL), TSH (mIU/L), SHBG (nmol/L).
Modifications in body composition | From baseline through study completion, estimated to be in 2035.
  Describe, in AFAB and AMAB transgender individuals who have been receiving gender-affirming hormone therapy (GAHT) for at least one year, changes in the following indicators of cardiovascular health: Body composition (DXA): Change in fat mass (kg), body-fat % (%), lean mass (kg), lean mass + BMC (kg), total body mass (kg).
Changes in insulin resistance | From baseline through study completion, estimated to be in 2035.
  Describe, in AFAB and AMAB transgender individuals who have been receiving gender-affirming hormone therapy (GAHT) for at least one year, changes in the following indicators of cardiovascular health: Insulin resistance indices: HOMA-IR (unitless), TyG index (unitless).

SECONDARY OUTCOMES:
Presence/absence of cardiovascular disease | From baseline through study completion, estimated to be in 2035.
  Calculate the incidence of conditions that increase cardiovascular risk-such as diabetes mellitus, arterial hypertension, hypercholesterolemia, hypertriglyceridemia, hepatic steatosis, and similar disorders-and determine whether specific medical treatments are required or whether gender-affirming hormone therapy should be discontinued.
Lifestyle habits of transgender individuals | From baseline through study completion, estimated to be in 2035.
  Describe the lifestyle-including diet, physical activity, and related factors-in AFAB and AMAB transgender individuals undergoing gender-affirming hormone therapy. Specifically, the study will evaluate the following variables: smoking, quantified in pack-years; alcohol intake, reported as the number of standard alcohol units; use of other substances, recorded as present or absent based on participant self-report; physical activity, calculated using the Exercise Vital Sign metric; and dietary pattern, self-reported as unrestricted, vegetarian, vegan, ketogenic, or another specified regimen.
Changes in cardiovascular health parameters according to the various types of GAHT | From baseline through study completion, estimated to be in 2035.
  Describe the changes in cardiovascular health parameters according to the type of gender-affirming hormone therapy administered-namely, transdermal testosterone versus injectable testosterone esters, or transdermal estradiol versus oral estradiol valerate combined with an anti-androgen.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual data will be shared anonymously upon reasonable request to the Principal Investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR